CLINICAL TRIAL: NCT02986958
Title: Involving Family to Improve Primary Care Visits for Cognitively Impaired Patients
Brief Title: Involving Family to Improve Communication in Primary Care
Acronym: SAMEPage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Johns Hopkins Community Physicians (Other); Medstar Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: R21AG049967 (NIH)
Record Dates: First submitted 2016-12-06; First posted 2016-12-08 (Estimated); Results first posted 2018-10-11 (Actual); Last update posted 2018-12-31 (Actual); Status verified 2018-12

CONDITIONS: Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Checklist (Experimental): One-page paper-pencil agenda setting checklist involving two activities for older primary care patients and their family companion. The purpose of the checklist is to 1. clarify the role of the family companion during the visit, and 2. to discuss patient health issues to discuss with the primary care provider
  Interventions: Other: Pre-visit patient-family agenda-setting checklist
- Usual Care (Placebo Comparator): Care as usual with their primary care provider
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Pre-visit patient-family agenda-setting checklist — Pre-visit patient-family agenda-setting checklist
  Arms: Checklist
Other: Usual care — routine primary care
  Arms: Usual Care

SUMMARY:
This study evaluates an agenda-setting checklist for patients with cognitive impairment and their family companions that is completed in the waiting room in advance of a primary care visit. The study team will conduct a two-group randomized trial to examine feasibility of the protocol and to compare medical communication (from visit audiotapes) during visits of patient-companion dyads who complete the checklist (n=50) with patient-companion dyads who receive usual care (n=50)

DETAILED DESCRIPTION:
The study team has established proof of concept for a paper-pencil checklist to be used by older patients and their companions in the waiting room prior to medical visits. The checklist is designed to elicit and align patient and companion perspectives regarding patient health issues to discuss with the doctor, and to stimulate discussion about the companion's role in the visit. The premise for the checklist is that companions are typically motivated to support patients during medical visits, but that they often lack knowledge of the patient's health concerns and preferences for communication assistance.

The study team will conduct a two group pilot randomized trial of up to 100 (50 per group) patients ages 65+ with cognitive impairment and their unpaid companion to test the effects of the refined checklist for medical communication. Each patient-companion dyad will be randomized to the intervention (to receive the checklist) or to a control protocol. The study will evaluate the feasibility of delivering the study protocol to patients with cognitive impairment and their companions in primary care, and to generate preliminary evidence regarding the effect of the checklist on medical communication. For these reasons, the control group protocol will comprise usual care which is in this case existing clinical practice. Patients (when feasible), companions, and doctors in both intervention and control groups will complete in-person post-visit surveys immediately after the visit. Patients (when feasible) and companions will separately complete follow-up surveys by telephone two weeks after the doctor visit conducted by a research staff member.

ELIGIBILITY:
Inclusion Criteria:

* Older adults: 65 years or older, established patient of participating primary care provider, regularly attend medical visits with one or more family member or unpaid friend "companion(s)", agree to allow companion to be contacted and participate in the study, authorize disclosure of Protected Health Information (PHI) in their electronic health record, able to provide informed consent or have a legally authorized representative
* Companion: family member (spouse, adult child, parent, adult sibling) or unpaid friend who accompanies older adult participant to medical visits.
* Primary care provider: practicing physician, nurse practitioner or physician assistant at a participating primary care practice.

Exclusion Criteria:

* Older adults: younger than 65 years, no evidence of cognitive impairment, do not attend medical visits with family member or unpaid friend.
* Companion: paid non-family member who accompanies patient to visits

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 93 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Wolff, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (3):
- United States (3):
  - Johns Hopkins Community Physicians, Aberdeen, Maryland
  - Medstar Center for Successful Aging, Baltimore, Maryland
  - Johns Hopkins Community Physicians, Westminster, Maryland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wolff JL, Roter DL, Barron J, Boyd CM, Leff B, Finucane TE, Gallo JJ, Rabins PV, Roth DL, Gitlin LN. A tool to strengthen the older patient-companion partnership in primary care: results from a pilot study. J Am Geriatr Soc. 2014 Feb;62(2):312-9. doi: 10.1111/jgs.12639. Epub 2014 Jan 13. PMID 24417565
- [Background] Wolff JL, Guan Y, Boyd CM, Vick J, Amjad H, Roth DL, Gitlin LN, Roter DL. Examining the context and helpfulness of family companion contributions to older adults' primary care visits. Patient Educ Couns. 2017 Mar;100(3):487-494. doi: 10.1016/j.pec.2016.10.022. Epub 2016 Oct 25. PMID 27817986
- [Derived] Wolff JL, Roter DL, Boyd CM, Roth DL, Echavarria DM, Aufill J, Vick JB, Gitlin LN. Patient-Family Agenda Setting for Primary Care Patients with Cognitive Impairment: the SAME Page Trial. J Gen Intern Med. 2018 Sep;33(9):1478-1486. doi: 10.1007/s11606-018-4563-y. Epub 2018 Jul 18. PMID 30022409

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Checklist | Usual Care
Started | 49 | 44
Completed | 49 | 44
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Checklist | Usual Care | Total
Number analyzed (Participants) | 49 | 44 | 93
Age, Continuous [Mean (Standard Deviation); unit: years] | 80.9 (8.0) | 78.8 (7.1) | 79.9 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 24 | 48
  Male | 25 | 20 | 45
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Nonwhite race or Hispanic ethnicity | 18 | 21 | 39
Mean Mini-Mental State Examination (MMSE) [Mean (Standard Deviation); unit: units on a scale] — The Mini-Mental State Examination (MMSE) is a 30-item questionnaire used to measure cognitive impairment in clinical and research settings. MMSE scores range from 0-30, with higher values indicating less impairment.
  units on a scale | 20.8 (7.8) | 22.5 (5.5) | 21.6 (6.8)

OUTCOME MEASURES:

1. Primary Outcome: Ratio of Psychosocial and Socio-emotional Statements Relative to Biomedical Talk and Orientation Statements (Patient-Centered Communication)
Description: Patient-centered communication is reflected as a ratio of psychosocial and socio-emotional statements relative to biomedical talk and orientation statements from coded audio-taped communication during primary care visits. Higher values indicate more patient-centered communication.
Time Frame: During enrollment visit, up to 77 minutes
Measure: Mean (Standard Error); unit: Ratio
Arm/Group | Checklist | Usual Care
Number analyzed (Participants) | 49 | 44
Ratio | 0.86 (0.42) | 0.68 (0.45)
Statistical Analysis 1: Comparison: Checklist vs Usual Care; Test type: Other — We used generalized estimating equations with an exchangeable correlation structure to assess the direction, magnitude, and statistical significance of between-group differences. Regression models included treatment assignment and patient-level covariates (patient age, gender, and MMSE score) that were postulated as affecting communication outcomes. Statistical tests were 2-sided with a significance level of 0.05. Analyses were performed in SAS statistical software, version 9.4 (SAS, Cary, NC); p = 0.046, t-test, 2 sided; Mean Difference (Final Values) = 0.16, Standard Error of Mean 0.08

2. Secondary Outcome: Visit Duration
Description: Duration of primary care visit in minutes
Time Frame: During enrollment visit, up to 77 minutes
Measure: Mean (Standard Error); unit: minutes
Arm/Group | Checklist | Usual Care
Number analyzed (Participants) | 49 | 44
minutes | 25.5 (12.5) | 24.8 (15.2)

3. Secondary Outcome: Patient Verbal Activity
Description: Patient verbal activity is the proportion of visit statements contributed by the patient in relation to overall visit statements, including statements by the companion and primary care provider.
Time Frame: During enrollment visit, up to 77 minutes
Measure: Mean (Standard Error); unit: Proportion of visit statements
Arm/Group | Checklist | Usual Care
Number analyzed (Participants) | 49 | 44
Proportion of visit statements | .226 (0.14) | .271 (0.14)

4. Secondary Outcome: Companion Verbal Activity
Description: Companion verbal activity is the proportion of visit statements contributed by the companion in relation to overall visit statements, including statements by the patient and primary care provider.
Time Frame: During enrollment visit, up to 77 minutes
Measure: Mean (Standard Error); unit: Proportion of visit statements
Arm/Group | Checklist | Usual Care
Number analyzed (Participants) | 49 | 44
Proportion of visit statements | .228 (0.14) | .182 (0.12)

5. Secondary Outcome: Number of Participants for Whom There Was Any Discussion of the Patient's Memory and/or Cognition During the Primary Care Visit
Description: The number of participants for whom there was any discussion of the patient's memory and/or cognition during the audio-recorded primary care visit.
Time Frame: During enrollment visit, up to 77 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Checklist | Usual Care
Number analyzed (Participants) | 49 | 44
Participants | 17 | 16

6. Secondary Outcome: Number of Patients Who Agree or Strongly Agree With Being Satisfied With the Primary Care Visit
Description: The number of patients who endorsed "Agree" or "Strongly Agree" to the statement: "Overall, I was satisfied with today's visit."
Time Frame: During Enrollment visit, up to 77 minutes
Population: The number of patient participants for this patient-reported outcome measure sums to 86 because 7 of the 93 total patient participants were too cognitively impaired to respond to the paper-pencil post-visit survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Checklist | Usual Care
Number analyzed (Participants) | 43 | 43
Participants | 43 | 43

7. Secondary Outcome: Number of Companions Who Agree or Strongly Agree With Being Satisfied With the Primary Care Visit
Description: The number of companions who endorsed "Agree" or "Strongly Agree" to the statement: "Overall, I was satisfied with today's visit."
Time Frame: During Enrollment visit, up to 77 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Checklist | Usual Care
Number analyzed (Participants) | 49 | 44
Participants | 49 | 44

8. Secondary Outcome: Number of Primary Care Providers Who Agree or Strongly Agree With Being Satisfied With the Primary Care Visit
Description: The number of primary care providers who endorsed "Agree" or "Strongly Agree" to the statement: "Overall, I was satisfied with today's visit."
Time Frame: During Enrollment visit, up to 77 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Checklist | Usual Care
Number analyzed (Participants) | 49 | 43
Participants | 46 | 43

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Checklist | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/44
Other Adverse Events (participants affected / at risk) | 0/49 | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-24): https://cdn.clinicaltrials.gov/large-docs/58/NCT02986958/Prot_SAP_000.pdf